CLINICAL TRIAL: NCT06443957
Title: The Preventive Effect and Safety of Different Doses of Insulin Nasal Administration on Postoperative Delirium in Elderly Hip Fracture Patients - a Randomized, Single Blind, Parallel Controlled, Single Center Clinical Trial
Brief Title: The Preventive Effect of Different Doses of Intranasal Insulin on Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23K214-001
Record Dates: First submitted 2024-05-07; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; Insulin; Intranasal administration
MeSH Terms: conditions — Emergence Delirium; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intranasal normal saline (Placebo Comparator): The patient was given 1ml of normal saline intranasally at 19:00 on the first day of surgery, 50 minutes before anesthesia on the day of surgery, and 19:00 on the day of surgery.
  Interventions: Drug: Intranasal normal saline
- Intranasal insulin-20U (Experimental): The patient was given 1ml of 20U insulin intranasally at 19:00 on the first day of surgery, 50 minutes before anesthesia on the day of surgery, and 19:00 on the day of surgery.
  Interventions: Drug: Intranasal insulin-20U
- Intranasal insulin-40U (Experimental): The patient was given 1ml of 40U insulin intranasally at 19:00 on the first day of surgery, 50 minutes before anesthesia on the day of surgery, and 19:00 on the day of surgery.
  Interventions: Drug: Intranasal insulin-40U

INTERVENTIONS:
Drug: Intranasal normal saline — The patient was given 1ml of normal saline intranasally at 19:00 on the first day of surgery, 50 minutes before anesthesia on the day of surgery, and 19:00 on the day of surgery.
  Arms: Intranasal normal saline
Drug: Intranasal insulin-20U — The patient was given 1ml of 20U insulin intranasally at 19:00 on the first day of surgery, 50 minutes before anesthesia on the day of surgery, and 19:00 on the day of surgery.
  Arms: Intranasal insulin-20U
Drug: Intranasal insulin-40U — The patient was given 1ml of 40U insulin intranasally at 19:00 on the first day of surgery, 50 minutes before anesthesia on the day of surgery, and 19:00 on the day of surgery.
  Arms: Intranasal insulin-40U

SUMMARY:
Postoperative delirium is one of the common complications in the older aldults after surgery, which can lead to longer hospita stay，memory loss and reduced quality of life. There is currently no specific treatment. Therefore, it is important to prevent the occurrence of postoperative delirium. This study investigated the effect of intranasal insulin administration on the prevention of postoperative delirium and compared different doses of insulin to find a safe and acceptable method for preventing delirium.

DETAILED DESCRIPTION:
Hip fractures are a common trauma in older adults and occur mainly in older people with osteoporosis. Surgery is the preferred choice for the vast majority of patients with severe pain and limited mobility in older aldults with hip fractures, resulting in higher mortality and disability rates with conservative treatment. But postoperative delirium becomes a challenge. At present, the treatment of delirium includes pharmacological and non-pharmacological methods, but the effect is limited, and now the focus is on preventing delirium, so this study investigated the effect of intranasal insulin administration on the prevention of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

Patients with hip fracture scheduled for unilateral hip arthroplasty or intramedullary nailing under subarachnoid block.

Both genders. Age ≥65 years old. Body mass index (BMI) ≤24kg/m2. American Society of Anesthesiologists (ASA) grade I-III.

Exclusion Criteria:

Contraindications to nasal administration (nasal defects or lesions). History of insulin allergy. Inability to communicate preoperatively (coma, severe visual or hearing impairment).

History of severe heart,Liver and kidney disease. History of psychiatric disorders. Preoperative delirium. Multiple traumas or fractures. Contraindications to subarachnoid block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

PRIMARY OUTCOMES:
postoperative delirium | From 18:00 to 19:00 on the 1st postoperative day, the 2nd postoperative day, and the 3rd postoperative day,
  The CAM-ICU scale is used to evaluate whether postoperative delirium occurs in three groups of patients. The scale is divided into four parts: acute changes and fluctuations in consciousness state, attention disorders, changes in consciousness level, and cognitive confusion. If acute changes in consciousness and attention deficit occur simultaneously, combined with changes in consciousness level and cognitive confusion, either can be diagnosed as postoperative delirium.

SECONDARY OUTCOMES:
visual analogue scale | On the 1st postoperative day, the 2nd postoperative day, and the 3rd postoperative day,
  Assess postoperative pain，0 represents painless, 10 represents severe pain, and the higher the score, the more severe the pain will be.
Lactate content in cerebrospinal fluid | During the anesthesia
  The patient underwent neuraxial anesthesia to obtain 0.5ml of cerebrospinal fluid and measure the lactate content in the cerebrospinal fluid
Blood glucose values | 1 day before the operation, 40 minutes after nasal administration of insulin or normal saline, before surgery and immediately after surgery
  A blood glucose meter is used to measure the patient's fingerstick blood glucose
Glucose content in cerebrospinal fluid | During the anesthesia
  The patient underwent neuraxial anesthesia to obtain 0.5ml of cerebrospinal fluid and measure the glucose content in the cerebrospinal fluid

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, China

REFERENCES:
- [Result] Marcantonio ER. Delirium in Hospitalized Older Adults. N Engl J Med. 2017 Oct 12;377(15):1456-1466. doi: 10.1056/NEJMcp1605501. PMID 29020579
- [Result] Oh ES, Fong TG, Hshieh TT, Inouye SK. Delirium in Older Persons: Advances in Diagnosis and Treatment. JAMA. 2017 Sep 26;318(12):1161-1174. doi: 10.1001/jama.2017.12067. PMID 28973626
- [Result] Craft S, Raman R, Chow TW, Rafii MS, Sun CK, Rissman RA, Donohue MC, Brewer JB, Jenkins C, Harless K, Gessert D, Aisen PS. Safety, Efficacy, and Feasibility of Intranasal Insulin for the Treatment of Mild Cognitive Impairment and Alzheimer Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2020 Sep 1;77(9):1099-1109. doi: 10.1001/jamaneurol.2020.1840. PMID 32568367
- [Result] Huang Q, Li Q, Qin F, Yuan L, Lu Z, Nie H, Gong G. Repeated Preoperative Intranasal Administration of Insulin Decreases the Incidence of Postoperative Delirium in Elderly Patients Undergoing Laparoscopic Radical Gastrointestinal Surgery: A Randomized, Placebo-Controlled, Double-Blinded Clinical Study. Am J Geriatr Psychiatry. 2021 Dec;29(12):1202-1211. doi: 10.1016/j.jagp.2021.02.043. Epub 2021 Feb 23. PMID 33757723
- [Derived] Li Y, Zhang Y, Ren Y, Liu H. Optimal Dose of Intranasal Insulin Administration for Reducing Postoperative Delirium Incidence in Older Patients Undergoing Hip Fracture Surgery. Am J Geriatr Psychiatry. 2025 Aug;33(8):891-900. doi: 10.1016/j.jagp.2025.03.009. Epub 2025 Mar 21. PMID 40222886